CLINICAL TRIAL: NCT03481972
Title: A Phase III Randomized Study of Doxycycline and Tauroursodeoxycholic Acid (Doxy/TUDCA) Plus Standard Supportive Therapy Versus Standard Supportive Therapy Alone in Cardiac Amyloidosis Caused by Transthyretin
Brief Title: A Study of Doxycycline and Tauroursodeoxycholic Acid (Doxy/TUDCA) Plus Standard Supportive Therapy Versus Standard Supportive Therapy Alone in Cardiac Amyloidosis Caused by Transthyretin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Giovanni Palladini, Professor, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC 011 IT
Record Dates: First submitted 2018-03-16; First posted 2018-03-29 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: TTR Cardiac Amyloidosis
MeSH Terms: interventions — Doxycycline; ursodoxicoltaurine; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doxy/TUDCA (Experimental): doxycicline (100 mg / BID)
  tauroursodeoxycholic acid (250 mg / TID)
  Interventions: Drug: Doxycycline and tauroursodeoxycholic acid
- Standard of care (Active Comparator): Standard of care therapies.
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Doxycycline and tauroursodeoxycholic acid — doxycicline and tauroursodeoxycholic acid
  Other Names: Standard of care therpay
  Arms: Doxy/TUDCA
Drug: Standard of care — Standard of care
  Arms: Standard of care

SUMMARY:
Cardiac amyloidosis caused by transthyretin either mutated (in ATTRm amyloidosis) or wildtype (in ATTRwt, formerly senile, amyloidosis) is a rare disease but is diagnosed with increasing frequency thanks to the availability of non-invasive scintigraphy-based means. Cardiac ATTR amyloidosis is characterized by progressive heart failure with a median survival of less than 4 years, and there is no standard treatment for this disease. It was proved that the marketed antibiotic doxycycline (Doxy) disrupts amyloid fibrils in vitro and in animal models synergistically with tauroursodeoxycholic acid (TUDCA). Based on these pre-clinical data, a clinical trial of Doxy/TUDCA in ATTR Amyloidosis (NCT01171859) was conducted.

Treatment was well tolerated and was able to prevent progression of cardiac dysfunction.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria:

* Diagnosis of ATTRwt amyloidosis, or ATTRm p.Ile68Leu and p.Val122Ile;
* the diagnosis of amyloidosis needs to be biopsy-proven, and amyloid deposits need to be characterized as ATTR-type by immuno-electron microscopy or mass spectrometry. Biopsy can be omitted in patients with a positive (score 3) cardiac 99mTc-DPD scintigraphy, provided serum and urine immunofixation does not show monoclonal components. Wild-type and mutated ATTR amyloidosis will be differentiated by DNA analysis;
* 18 years or older;
* cardiac involvement (mean left ventricular wall thickness >12 mm in the absence of other causes);
* history of occurrence of at least 1 event of symptomatic heart failure;
* stable diuretic dosage for at least 2 weeks before treatment initiation;
* female patients who are postmenopausal for at least 1 year before the screening visit, or are surgically sterile, or if they are of childbearing potential, agree to practice effective methods of contraception from the time of signing the informed consent through 30 days after the last dose of study drug, or agree to completely abstain from intercourse;
* voluntary written consent must be given before performance of any study-related procedure not part of standard medical care with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

Exclusion Criteria:

Subjects must meet none of the following criteria:

* Non-ATTR amyloidosis;
* NYHA class IV;
* enzyme-documented myocardial infarction within 6 months before enrollment;
* pregnant or nursing women;
* uncontrolled bacterial, viral, fungal, HIV, HBV, or HCV infection;
* presence of other active malignancy with the exception of non-melanoma skin cancer, cervical cancer, treated early-stage prostate cancer provided that prostate specific antigen is within normal limit, or any completely resected carcinoma in situ;
* known allergy to any of the study medications, their analogues, or excipients in the various formulations;
* treatment with drugs potentially affecting doxycycline absorption;
* significant acute gastrointestinal symptoms;
* active peptic ulceration and/or esophageal reflux disease;
* treatment with any investigational products within 28 days before the first dose of study drug;
* requirement for other concomitant chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered to be investigational;
* any other serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
evaluate the efficacy of Doxy/TUDCA in patients with cardiac ATTR amyloidosis, comparing survival free at 18 months of patients receiving Doxy/TUDCA + standard supportive therapy with that of patients in standard supportive therapy alone. | 18 MONTHS
  Doxy/TUDCA efficacy

SECONDARY OUTCOMES:
Compare overall survival at 18 and 30 months of patients receiving Doxy/TUDCA in addition to standard supportive therapy with that of patients receiving standard supportive therapy alone. | 18 and 30 months
  Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy